CLINICAL TRIAL: NCT05689229
Title: Aerosolized Versus Intravenous Colistin-based Antimicrobial Regimens in Hospitalized COVID-19 Patients With Bacterial Coinfection: A Randomized Controlled Trial
Acronym: colistin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Clinical Pharmacy Department, Faculty of Pharmacy, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSU-22006
Record Dates: First submitted 2023-01-13; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Secondary Bacterial Infection in COVID-19 Patients
MeSH Terms: interventions — Colistin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colistin IV (Active Comparator)
  Interventions: Drug: Colistin
- Colistin Aerosolized (Active Comparator)
  Interventions: Drug: Colistin
- Control (No Intervention)

INTERVENTIONS:
Drug: Colistin — COVID-19 patients with secondary gram-negative bacterial infections receive colistin IV or aerosolized
  Arms: Colistin Aerosolized; Colistin IV

SUMMARY:
Secondary bacterial pathogen infection has been demonstrated to aggravate COVID-19 clinical outcomes. Bacterial infections acquired during a hospital stay are likely resistant to several antimicrobial medicines, making COVID-19 patient management difficult. As a result, it is believed that aerosolized colistin might be a viable choice for treating secondary bacterial infections caused by gram-negative resistant strains in individuals who also have COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 patients with secondary gram-negative bacterial infections

Exclusion Criteria:

* Patients with resistant bacterial strains to polymyxins
* patients less than 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Microbial eradication | 10 days
Mortality | 30 days

SECONDARY OUTCOMES:
Nephrotoxicity | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt